CLINICAL TRIAL: NCT00613327
Title: The Efficacy of Oxybutynin Chloride OROS in Patient-Reported Outcomes With Dose Escalation in Korean Overactive Bladder Patients
Brief Title: An Efficacy and Safety Study of Oxybutynin Chloride Oral Osmotic Therapeutic System (OROS) in Korean Overactive Bladder Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013840; OXY-KOR-4001
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2013-09-16 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-10

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive bladder; Oxybutynin chloride; OROS
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxybutynin Chloride OROS (Experimental)
  Interventions: Drug: Oxybutynin chloride OROS

INTERVENTIONS:
Drug: Oxybutynin chloride OROS — Participants will receive oxybutynin chloride OROS tablet at starting dose of 10 milligram (mg) orally once daily. The dose will be adjusted by 10 mg every 2 weeks up to first 6 weeks, based on the criteria for evaluation of optimal dose. The optimal dose obtained in first 6 weeks will be continued up to Week 12. Maximum allowed dose will be 30 mg per day.
  Other Names: Lyrinel

SUMMARY:
The objective of this study is to evaluate the efficacy of oxybutynin chloride oral osmotic therapeutic system (OROS) on patient-reported outcomes after 12 weeks of treatment by dose escalation in participants with overactive bladder.

DETAILED DESCRIPTION:
This is a multicenter (when more than one hospital or medical school team work on a medical research study), open-label (all people know the identity of the intervention), prospective (study following participants forward in time) Phase 4 study of oxybutynin chloride OROS in participants with overactive bladder. The total study duration will be 12 weeks and will include following visits: Screening (Week -2), Baseline, Week 2, 4, 6 and 12. Participants will receive oxybutynin chloride OROS tablet at starting dose of 10 milligram (mg) orally once daily. The dose will be adjusted by 10 mg every 2 weeks up to first 6 weeks, based on the criteria for evaluation of optimal dose. The optimal dose obtained in first 6 weeks will be continued up to Week 12. Maximum allowed dose will be 30 mg per day. Efficacy will primarily be evaluated by assessment of goal achievement (percentage of participants who show a score 4 or 5 in the Likert scale for treatment goal) at Week 12. Participants' safety will also be monitored at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants who fulfilled all of the following criteria in their micturition charts completed for 3 days prior to visit 2 (Baseline): mean voiding frequency greater than or equal to 8 times per 24 hours and mean frequency of urinary urgency greater than or equal to 2 times per 24 hours (urgency means sudden and strong urge to urinate and a urinary sensation scale score greater than or equal to 3 in the micturition chart)
* Participants with overactive bladder symptoms lasting for 3 months or longer prior to study initiation
* Participants who were capable of completing micturition chart and survey questionnaires and provided informed consent to complete them
* Participants who could sign on the informed consent form after fully listening to and understanding about characteristics, risks and benefits of the study

Exclusion Criteria:

* Participants with stress urinary incontinence (not able to control bladder actions) or participants with complicated incontinence dominantly presenting stress urinary incontinence when judging based on medical history
* Participants with a hepatic (pertaining to liver) or renal (pertaining to kidneys) disease indicating serum aspartate transaminase (AST [SGOT]), alanine transaminase (ALT [SGPT]), alkaline phosphatase or creatinnine concentration twice or more of normal upper limit
* Participants contraindicated to use anticholinergics including uncontrolled narrow angle glaucoma (increased pressure inside the eye that causes visual problems), urinary retention or gastrointestinal tract retention
* Participants experiencing a symptom of acute urinary tract infection (UTI) during the run-in period
* Participants with recurrent UTI who had medical history of treatment for UTI symptom 5 times or more in the past one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxybutynin Chloride OROS: Oxybutynin chloride osmotic release oral system (OROS) tablet at starting dose of 10 milligram (mg) orally once daily. The dose was adjusted by 10 mg every 2 weeks up to first 6 weeks, based on the criteria for evaluation of optimal dose. The optimal dose obtained in first 6 weeks was continued up to Week 12. Maximum allowed dose was 30 mg per day.
Period: Overall Study
Arm/Group | Oxybutynin Chloride OROS
Started | 345
Completed | 244
Not Completed | 101
Not completed — Adverse Event | 38
Not completed — Lost to Follow-up | 8
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 2
Not completed — Other | 47

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who received study drug at least once and had data for efficacy evaluation (goal achievement in treatment) available.
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 309
Age Continuous [Mean (Standard Deviation); unit: Years] | 54.93 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 256
  Male | 53

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Treatment Goal
Description: Goal achievement was measured by using the 6-point Likert scale (0=not achieved at all and 5=completely achieved). Achievement of treatment goal was defined by a score of 4 or 5 in the Likert scale. Percentage of participants who achieved their treatment goal defined at Baseline (for a maximum of 3 items among the 10 items including incontinence, urinary urgency, frequent urination, nocturnal frequent urination, tenesmus, general health, life habit, activity, pain/pressure pain, and sexual function) was reported.
Time Frame: Week 12
Population: ITT population included all participants who received study drug at least once and had data for efficacy evaluation (goal achievement in treatment) available. Missing data at Week 12 were imputed using last observation carried forward (LOCF).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 309
Percentage of participants | 40.45 [34.93 to 46.16]

2. Secondary Outcome: Number of Participants With Change From Baseline in Response to Primary Overactive Bladder (OAB) Symptom Questionnaire (POSQ): Urinary Urgency at Week 12
Description: Participants assessed their bothering for overactive bladder symptom by completing POSQ rated on a 5-point scale: how much they were bothered by urinary urgency (strong micturition desire indicated) in the past two weeks. The responses were indicated as: 1 (not bothered at all), 2 (slightly bothered), 3 (average), 4 (strongly bothered) and 5 (very strongly bothered). Number of participants with change from Baseline in the response to this question at Week 12 was reported.
Time Frame: Baseline and Week 12
Population: ITT population included all participants who received study drug at least once and had data for efficacy evaluation (goal achievement in treatment) available. Here 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Participants
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 275
Participants
  Baseline: Not bothered, Week 12: Not bothered | 1
  Baseline: Not bothered, Week 12: Slightly | 2
  Baseline: Not bothered, Week 12: Average | 0
  Baseline: Not bothered, Week 12: Strongly | 0
  Baseline: Not bothered, Week 12: Very strongly | 0
  Baseline: Slightly, Week 12: Not bothered | 17
  Baseline: Slightly, Week 12: Slightly | 29
  Baseline: Slightly, Week 12: Average | 12
  Baseline: Slightly, Week 12: Strongly | 6
  Baseline: Slightly, Week 12: Very strongly | 1
  Baseline: Average, Week 12: Not bothered | 13
  Baseline: Average, Week 12: Slightly | 22
  Baseline: Average, Week 12: Average | 17
  Baseline: Average, Week 12: Strongly | 2
  Baseline: Average, Week 12: Very strongly | 0
  Baseline: Strongly, Week 12: Not bothered | 18
  Baseline: Strongly, Week 12: Slightly | 41
  Baseline: Strongly, Week 12: Average | 40
  Baseline: Strongly, Week 12: Strongly | 16
  Baseline: Strongly, Week 12: Very strongly | 5
  Baseline: Very strongly, Week 12: Not bothered | 5
  Baseline: Very strongly, Week 12: Slightly | 14
  Baseline: Very strongly, Week 12: Average | 4
  Baseline: Very strongly, Week 12: Strongly | 4
  Baseline: Very strongly, Week 12: Very strongly | 6

3. Secondary Outcome: Number of Participants With Change From Baseline in Response to Primary Overactive Bladder (OAB) Symptom Questionnaire (POSQ): Frequent Daytime Urination at Week 12
Description: Participants assessed their bothering for overactive bladder symptom by completing POSQ rated on a 5-point scale: how much they were bothered by daytime frequent urination (frequent urination was required more than the frequency desired during daytime) in the past two weeks. The responses were indicated as: 1 (not bothered at all), 2 (slightly bothered), 3 (average), 4 (strongly bothered) and 5 (very strongly bothered). Number of participants with change from Baseline in the response to this question at Week 12 was reported.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 275
Participants
  Baseline: Not bothered, Week 12: Not bothered | 3
  Baseline: Not bothered, Week 12: Slightly | 3
  Baseline: Not bothered, Week 12: Average | 0
  Baseline: Not bothered, Week 12: Strongly | 0
  Baseline: Not bothered, Week 12: Very strongly | 0
  Baseline: Slightly, Week 12: Not bothered | 7
  Baseline: Slightly, Week 12: Slightly | 15
  Baseline: Slightly, Week 12: Average | 10
  Baseline: Slightly, Week 12: Strongly | 2
  Baseline: Slightly, Week 12: Very strongly | 0
  Baseline: Average, Week 12: Not bothered | 19
  Baseline: Average, Week 12: Slightly | 22
  Baseline: Average, Week 12: Average | 21
  Baseline: Average, Week 12: Strongly | 6
  Baseline: Average, Week 12: Very strongly | 0
  Baseline: Strongly, Week 12: Not bothered | 21
  Baseline: Strongly, Week 12: Slightly | 36
  Baseline: Strongly, Week 12: Average | 36
  Baseline: Strongly, Week 12: Strongly | 22
  Baseline: Strongly, Week 12: Very strongly | 4
  Baseline: Very strongly, Week 12: Not bothered | 4
  Baseline: Very strongly, Week 12: Slightly | 17
  Baseline: Very strongly, Week 12: Average | 12
  Baseline: Very strongly, Week 12: Strongly | 12
  Baseline: Very strongly, Week 12: Very strongly | 3

4. Secondary Outcome: Number of Participants With Change From Baseline in Response to Primary Overactive Bladder (OAB) Symptom Questionnaire (POSQ): Frequent Nighttime Urination at Week 12
Description: Participants assessed their bothering for overactive bladder symptom by completing POSQ rated on a 5-point scale: how much they were bothered by nighttime frequent urination (waking up from sleep in order to void urine at nighttime [period from time of going to bed to time planned to wake up in the morning]) in the past two weeks. The responses were indicated as: 1 (not bothered at all), 2 (slightly bothered), 3 (average), 4 (strongly bothered) and 5 (very strongly bothered). Number of participants with change from Baseline in the response to this question at Week 12 was reported.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 276
Participants
  Baseline: Not bothered, Week 12: Not bothered | 15
  Baseline: Not bothered, Week 12: Slightly | 3
  Baseline: Not bothered, Week 12: Average | 1
  Baseline: Not bothered, Week 12: Strongly | 0
  Baseline: Not bothered, Week 12: Very strongly | 0
  Baseline: Slightly, Week 12: Not bothered | 18
  Baseline: Slightly, Week 12: Slightly | 22
  Baseline: Slightly, Week 12: Average | 8
  Baseline: Slightly, Week 12: Strongly | 0
  Baseline: Slightly, Week 12: Very strongly | 1
  Baseline: Average, Week 12: Not bothered | 17
  Baseline: Average, Week 12: Slightly | 24
  Baseline: Average, Week 12: Average | 22
  Baseline: Average, Week 12: Strongly | 2
  Baseline: Average, Week 12: Very strongly | 0
  Baseline: Strongly, Week 12: Not bothered | 16
  Baseline: Strongly, Week 12: Slightly | 32
  Baseline: Strongly, Week 12: Average | 23
  Baseline: Strongly, Week 12: Strongly | 18
  Baseline: Strongly, Week 12: Very strongly | 3
  Baseline: Very strongly, Week 12: Not bothered | 6
  Baseline: Very strongly, Week 12: Slightly | 23
  Baseline: Very strongly, Week 12: Average | 7
  Baseline: Very strongly, Week 12: Strongly | 11
  Baseline: Very strongly, Week 12: Very strongly | 4

5. Secondary Outcome: Number of Participants With Change From Baseline in Response to Primary Overactive Bladder (OAB) Symptom Questionnaire (POSQ): Urge Urinary Incontinence at Week 12
Description: Participants assessed their bothering for overactive bladder symptom by completing POSQ rated on a 5-point scale: how much they were bothered by urge urinary incontinence (involuntary voiding or urinary leakage due to sudden micturition desire, not by sneezing, coughing or laughing) in the past two weeks. The responses were indicated as: 1 (not bothered at all), 2 (slightly bothered), 3 (average), 4 (strongly bothered) and 5 (very strongly bothered). Number of participants with change from Baseline in the response to this question at Week 12 was reported.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 276
Participants
  Baseline: Not bothered, Week 12: Not bothered | 63
  Baseline: Not bothered, Week 12: Slightly | 7
  Baseline: Not bothered, Week 12: Average | 5
  Baseline: Not bothered, Week 12: Strongly | 3
  Baseline: Not bothered, Week 12: Very strongly | 3
  Baseline: Slightly, Week 12: Not bothered | 28
  Baseline: Slightly, Week 12: Slightly | 19
  Baseline: Slightly, Week 12: Average | 2
  Baseline: Slightly, Week 12: Strongly | 2
  Baseline: Slightly, Week 12: Very strongly | 1
  Baseline: Average, Week 12: Not bothered | 19
  Baseline: Average, Week 12: Slightly | 13
  Baseline: Average, Week 12: Average | 7
  Baseline: Average, Week 12: Strongly | 2
  Baseline: Average, Week 12: Very strongly | 0
  Baseline: Strongly, Week 12: Not bothered | 14
  Baseline: Strongly, Week 12: Slightly | 22
  Baseline: Strongly, Week 12: Average | 13
  Baseline: Strongly, Week 12: Strongly | 10
  Baseline: Strongly, Week 12: Very strongly | 1
  Baseline: Very strongly, Week 12: Not bothered | 15
  Baseline: Very strongly, Week 12: Slightly | 17
  Baseline: Very strongly, Week 12: Average | 4
  Baseline: Very strongly, Week 12: Strongly | 5
  Baseline: Very strongly, Week 12: Very strongly | 1

6. Secondary Outcome: Patient's Perception of Symptom Improvement (PPSI) Score for Overactive Bladder
Description: Participant's perception about decrease in the most bothering symptom of overactive bladder (defined at Baseline) was evaluated by using visual analogue scale (VAS) at Week 12. The total score range was 0 to 100 where 0=symptom disappeared and 100=symptom unchanged or worsened compared to Baseline.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 275
Units on a scale | 38.66 (29.73)

7. Secondary Outcome: Number of Participants With Response to Patient's Perception of Treatment Benefit (PPTB) Questionnaire
Description: The PPTB was used to assess participant's perception about treatment benefit and satisfaction of the study drug. Regarding benefit, participants indicated whether they had any benefit obtained from the treatment. If yes, then the participants indicated whether it was weak benefit or strong benefit. Regarding satisfaction, participants indicated whether they were satisfied with the treatment. If yes, then they indicated if the treatment was slightly satisfactory or very satisfactory. If no, then they indicated if the treatment was slightly unsatisfactory or very unsatisfactory.
Time Frame: Week 2, 4, 6 and 12
Population: ITT population included all participants who received study drug at least once and had data for efficacy evaluation (goal achievement in treatment) available. Here 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure and 'n' specifies those participants who were evaluable for specific categories.
Measure: Number; unit: Participants
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 303
Participants
  Benefit: Week 2, Weak benefit (n=303) | 184
  Benefit: Week 2, Strong benefit (n=303) | 45
  Benefit: Week 2, No benefit (n=303) | 73
  Benefit: Week 2, Missing (n=303) | 1
  Benefit: Week 4, Weak benefit (n=281) | 155
  Benefit: Week 4, Strong benefit (n=281) | 86
  Benefit: Week 4, No benefit (n=281) | 39
  Benefit: Week 4, Missing (n=281) | 1
  Benefit: Week 6, Weak benefit (n=252) | 135
  Benefit: Week 6, Strong benefit (n=252) | 97
  Benefit: Week 6, No benefit (n=252) | 19
  Benefit: Week 6, Missing (n=252) | 1
  Benefit: Week 12, Weak benefit (n=277) | 117
  Benefit: Week 12, Strong benefit (n=277) | 127
  Benefit: Week 12, No benefit (n=277) | 32
  Benefit: Week 12, Missing (n=277) | 1
  Satisfaction: Week 2,Slightly satisfactory(n=302) | 168
  Satisfaction: Week 2,Very satisfactory(n=302) | 27
  Satisfaction:Week 2,Slightly unsatisfactory(n=302) | 52
  Satisfaction: Week 2, Very unsatisfactory (n=302) | 55
  Satisfaction: Week 4,Slightly satisfactory(n=282) | 160
  Satisfaction: Week 4, Very satisfactory (n=282) | 57
  Satisfaction:Week 4,Slightly unsatisfactory(n=282) | 37
  Satisfaction: Week 4, Very unsatisfactory (n=282) | 26
  Satisfaction: Week 4, Missing (n=282) | 2
  Satisfaction: Week 6,Slightly satisfactory(n=251) | 140
  Satisfaction: Week 6, Very satisfactory (n=251) | 68
  Satisfaction:Week 6,Slightly unsatisfactory(n=251) | 23
  Satisfaction: Week 6, Very unsatisfactory (n=251) | 19
  Satisfaction: Week 6, Missing (n=251) | 1
  Satisfaction: Week 12,Slightly satisfactory(n=277) | 136
  Satisfaction: Week 12, Very satisfactory (n=277) | 87
  Satisfaction:Week12,Slightly unsatisfactory(n=277) | 19
  Satisfaction: Week 12, Very unsatisfactory (n=277) | 34
  Satisfaction: Week 12, Missing (n=277) | 1

8. Secondary Outcome: Number of Participants With Response to Patient's Perception of Bladder Condition (PPBC) Questionnaire
Description: Participant's perception about bladder condition was evaluated by using self administered PPBC questionnaire. Participants answered "Which of the following statements describes your bladder condition best at the moment?" on a 6-point scale: 1= not problematic at all, 2=mild problem, 3=more or less a mild problem, 4=moderate problem, 5=severe problem and 6=very severe problem.
Time Frame: Baseline and Week 12
Population: ITT population included all participants who received study drug at least once and had data for efficacy evaluation (goal achievement in treatment) available. Here, 'n' specifies those participants who were evaluable for specific categories at given time point.
Measure: Number; unit: Participants
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 309
Participants
  Baseline: Not problematic at all (n=309) | 0
  Baseline: Mild problem (n=309) | 4
  Baseline: More or less a mild problem (n=309) | 25
  Baseline: Moderate problem (n=309) | 81
  Baseline: Severe problem (n=309) | 137
  Baseline:Very severe problem (n=309) | 62
  Week 12: Not problematic at all (n=275) | 20
  Week 12: Mild problem (n=275) | 66
  Week 12: More or less a mild problem (n=275) | 85
  Week 12: Moderate problem (n=275) | 63
  Week 12: Severe problem (n=275) | 30
  Week 12: Very severe problem (n=275) | 11

9. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire (OAB-q) Score at Week 6 and 12
Description: The OAB-q was used to evaluate influence of overactive bladder symptom on health-related quality of life (HRQL). It consisted of 2 parts: Symptom bother (6 items) evaluating how much symptoms related to overactive bladder were bothering in the last 4 weeks and HRQL (13 items) evaluating how general symptoms related to the bladder influenced life in the last 4 weeks. Each item was rated on 6-point Likert scale: 1 (not at all) to 6 (a very great deal). Total score range: 6 to 36 for symptom bother and 13 to 78 for HRQL. Transformed score calculated as ([Actual total raw score - lowest possible value of raw score]/range)*100 for symptom bother where higher score indicates greater symptom bother and as ([Highest possible raw score-Actual total raw score]/Raw score range)*100 for HRQL where higher scores indicate better HRQL. Transformed score range: 0-100 for both, symptom bother and HRQL.
Time Frame: Baseline, Week 6, 12 or early discontinuation (ED)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 309
Units on a scale
  Symptom bother: Baseline (n=309) | 50.08 (21.61)
  Symptom bother: Change at Week 6 (n=251) | -23.73 (22.63)
  Symptom bother: Change at Week 12/ED (n=276) | -25.63 (23.68)
  HRQL: Baseline (n=309) | 53.46 (21.20)
  HRQL: Change at Week 6 (n=251) | 18.96 (19.11)
  HRQL: Change at Week 12/ED (n=276) | 21.32 (22.01)

10. Secondary Outcome: Mean Voiding Frequency
Description: Mean voiding frequency for 24 hours was calculated as sum of total voiding frequency divided by the number of days when micturition chart was completed. Participants completed micturition chart for 3 days at Baseline, Week 6 and 12/ED. Mean daytime voiding frequency for 24 hours was calculated as sum of total daytime voiding frequency divided by the number of days when micturition chart was completed. Mean nighttime voiding frequency for 24 hours was calculated as sum of total nighttime voiding frequency divided by the number of days when micturition chart was completed. Nighttime voiding was defined as voiding during the sleep cycle.
Time Frame: Baseline, Week 6, 12 or ED
Population: ITT population included all participants who received study drug at least once and had data for efficacy evaluation (goal achievement in treatment) available. Here, 'n' specifies those participants who were evaluable for specific categories.
Measure: Mean (Standard Deviation); unit: Urinations per day
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 309
Urinations per day
  Daytime: Baseline (n=309) | 10.75 (3.71)
  Daytime: Week 6 (n=244) | 8.22 (2.78)
  Daytime: Week 12/ED (n=245) | 8.08 (3.55)
  Nighttime: Baseline (n=309) | 1.96 (1.75)
  Nighttime: Week 6 (n=244) | 1.34 (1.04)
  Nighttime: Week 12/ED (n=245) | 1.26 (1.40)
  Total: Baseline (n=309) | 12.71 (4.56)
  Total: Week 6 (n=244) | 9.56 (3.20)
  Total: Week 12/ED (n=245) | 9.34 (4.22)

11. Secondary Outcome: Percent Change From Baseline in Mean Voiding Frequency at Week 6 and 12
Description: Mean voiding frequency for 24 hours was calculated as sum of total voiding frequency divided by the number of days when micturition chart was completed. Participants completed micturition chart for 3 days at Baseline, Week 6 and 12/ED. Mean daytime voiding frequency for 24 hours was calculated as sum of total daytime voiding frequency divided by the number of days when micturition chart was completed. Mean nighttime voiding frequency for 24 hours was calculated as sum of total nighttime voiding frequency divided by the number of days when micturition chart was completed. Nighttime voiding was defined as voiding during the sleep cycle. Percent change was calculated as (change value/Baseline value)*100.
Time Frame: Baseline, Week 6, 12 or ED
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 309
Percent change
  Daytime: Percent change at Week 6 (n=244) | -20.36 (22.15)
  Daytime: Percent change at Week 12/ED (n=245) | -22.47 (25.76)
  Nighttime: Percent change at Week 6 (n=223) | -13.91 (80.74)
  Nighttime:Percent change at Week 12/ED (n=224) | -21.54 (80.72)
  Total: Percent change at Week 6 (n=244) | -22.19 (19.40)
  Total: Percent change at Week 12/ED (n=245) | -24.90 (22.06)

12. Secondary Outcome: Frequency of Urinary Urgency and Urinary Incontinence
Description: Urinary urgency means sudden and strong urge to urinate. It was rated by participant on 5-point scale (1=no urinary urgency and 5=urge urinary incontinence). Total frequency of urinary incontinence (UI) for 24 hours was calculated as sum of total frequency of incontinence divided by the number of days when micturition chart was completed. Participants completed micturition chart for 3 days at Baseline, Week 6 and 12/ED. Mean frequency of urinary urgency for 24 hours was calculated as sum of total frequency of urinary urgency divided by the number of days when micturition chart was completed. Urinary urgency was defined as voiding with urinary sensation scale score greater than or equal to 3.
Time Frame: Baseline, Week 6, 12 or ED
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Episodes per day
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 309
Episodes per day
  Urinary urgency: Baseline (n=309) | 9.40 (5.28)
  Urinary urgency: Week 6 (n=244) | 5.11 (4.25)
  Urinary urgency: Week 12/ED (n=245) | 4.31 (4.48)
  UI: Baseline (n=309) | 0.911 (3.244)
  UI: Week 6 (n=244) | 0.213 (0.959)
  UI: Week 12/ED (n=245) | 0.224 (1.203)

13. Secondary Outcome: Percent Change From Baseline in Frequency of Urinary Urgency and Urinary Incontinence at Week 6 and 12
Description: Urinary urgency means sudden and strong urge to urinate. It was rated by participant on 5-point scale (1=no urinary urgency and 5=urge urinary incontinence). Total frequency of UI for 24 hours was calculated as sum of total frequency of incontinence divided by the number of days when micturition chart was completed. Participants completed micturition chart for 3 days at Baseline, Week 6 and 12/ED. Mean frequency of urinary urgency for 24 hours was calculated as sum of total frequency of urinary urgency divided by the number of days when micturition chart was completed. Urinary urgency was defined as voiding with urinary sensation scale score greater than or equal to 3. Percent change was calculated as (change value/Baseline value)*100.
Time Frame: Baseline, Week 6, 12 or ED
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 309
Percent change
  Urinary urgency: Percent change at Week 6 (n=244) | -39.16 (72.56)
  Urinary urgency:Percent change at Week12/ED(n=245) | -46.19 (80.39)
  UI: Percent change at Week 6 (n=75) | -56.42 (107.15)
  UI: Percent change at Week 12/ED (n=75) | -74.64 (57.92)

14. Secondary Outcome: Mean Severity of Urinary Urgency at Urination
Description: Urinary urgency means sudden and strong urge to urinate. It was rated by participant on 5-point scale (1=no urinary urgency, 2=light urinary urgency, 3=moderate urinary urgency, 4=severe urinary urgency and 5=urge urinary incontinence). Mean severity of urinary urgency at urination was calculated as sum of all degrees of urinary urgency measured divided by the voiding frequency.
Time Frame: Baseline, Week 6, 12 or ED
Population: Data was reported in individual participant listings as planned, but not statistically summarized for analysis.
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 0

15. Secondary Outcome: Visual Analogue Scale (VAS) Score for Dry Mouth
Description: Severity of dry mouth was evaluated in participants by using VAS: how much dry mouth they have experienced in the past one week. The total score range was 0 (no dry mouth) to 100 (unimaginably most severe dry mouth).
Time Frame: Baseline, Week 6, 12 or ED
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 308
Units on a scale
  Baseline (n=308) | 20.30 (22.37)
  Week 6 (n=250) | 46.26 (26.46)
  Week 12/ED (n=277) | 43.85 (29.31)

16. Secondary Outcome: Percent Change From Baseline in Visual Analogue Scale (VAS) Score for Dry Mouth at Week 6 and 12
Description: Severity of dry mouth was evaluated in participants by using VAS: how much dry mouth they experienced in the past one week. The total score range was 0 (no dry mouth) to 100 (unimaginably most severe dry mouth). Percent change was calculated as (change value/Baseline value)*100.
Time Frame: Baseline, Week 6, 12 or ED
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Oxybutynin Chloride OROS
Number analyzed (Participants) | 308
Percent change
  Percent change at Week 6 (n=159) | 210.96 (701.21)
  Percent change at Week 12/ED (n=181) | 171.90 (475.90)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Description: Safety population included all participants who received the study drug at least once and had safety data available after starting the study treatment (N=320).
Arm/Group | Oxybutynin Chloride OROS
Serious Adverse Events (participants affected / at risk) | 3/320
Other Adverse Events (participants affected / at risk) | 289/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxybutynin Chloride OROS (N=320)
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Ventricular hypertrophy (Cardiac disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxybutynin Chloride OROS (N=320)
Dry mouth (Gastrointestinal disorders) | 261
Dyspepsia (Gastrointestinal disorders) | 33
Constipation (Gastrointestinal disorders) | 28
Gastrointestinal disorder (Gastrointestinal disorders) | 17
Diarrhoea (Gastrointestinal disorders) | 7
Abdominal discomfort (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Dysuria (Renal and urinary disorders) | 27
Urine flow decreased (Renal and urinary disorders) | 7
Urinary retention (Renal and urinary disorders) | 4
Bladder pain (Renal and urinary disorders) | 2
Urinary hesitation (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 2
Hypertonic bladder (Renal and urinary disorders) | 1
Pyuria (Renal and urinary disorders) | 1
Urethral pain (Renal and urinary disorders) | 1
Headache (Nervous system disorders) | 14
Somnolence (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Oedema (General disorders) | 8
Chest discomfort (General disorders) | 5
Face oedema (General disorders) | 4
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Dry eye (Eye disorders) | 6
Vision blurred (Eye disorders) | 4
Xerophthalmia (Eye disorders) | 2
Blepharospasm (Eye disorders) | 1
Cataract (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Nasopharyngitis (Infections and infestations) | 7
Acute sinusitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Prurigo (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 8
Insomnia (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No